CLINICAL TRIAL: NCT05247047
Title: A Post-market Cluster Randomized Controlled Trial of the Effect of the TENA SmartCare Change Indicator on Continence Care Efficiency and Skin Health in Long Term Care Facilities
Brief Title: The Effect of the TENA SmartCare Change Indicator on Care Efficiency and Skin Health in Long Term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WHEELS-ONE
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Cluster
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device (Experimental): Clusters in this arm will start using the device and use it for 6 weeks.
  Interventions: Device: TENA SmartCare Change Indicator
- Control (No Intervention): Clusters in this arm will not receive the device it will continue with usual care with no changes.

INTERVENTIONS:
Device: TENA SmartCare Change Indicator — The intervention is a medical device system that consists of a reusable electronic sensor and an application installed on one or more smart phones. The device estimates the saturation level of an absorbing incontinence product used by a study subject. The device is non-invasive and does not have any effect on the function of the absorbing incontinence product.
  Arms: Device

SUMMARY:
The purpose of this post market clinical investigation is to demonstrate the performance and safety of the TENA SmartCare Change Indicator when used in a nursing home setting.

DETAILED DESCRIPTION:
The TENA SmartCare Change Indicator is intended for use on individuals suffering from Urinary Incontinence who are cared for in a nursing home environment, by one or more professional caregivers. The TENA SmartCare Change Indicator is an accessory to TENA absorbing incontinence products. This clinical investigation is intended to demonstrate that use of TENA SmartCare Change Indicator has the ability to increase continence care efficiency at the nursing home by reducing the time needed in daily handling of absorbing incontinence products. Furthermore, this reduction in needed care does not have a detrimental effect on skin health. Secondarily, the investigation have multiple outcomes regarding number of checks, changes and leaks and also quality of life for subjects and qualitative measures for caregivers. Furthermore, the safety will continuously be monitored through analyzing device-related adverse events reported during the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has urinary incontinence managed with incontinence products with tapes, belted or pull up incontinence product type (products for moderate to heavy incontinence).
2. Subject is a permanent (intended length of stay four months or longer) resident of the nursing home.
3. Subject is unable to consistently communicate toileting needs.
4. Subject is unable to successfully toilet and change the pad without assistance.
5. Subject is using or is willing to use TENA Slip (Stretch) TENA Flex (Belted) and TENA Pants (Underwear) absorbing products for the study.
6. Subject has a waist size appropriate to the available sizes of incontinence products.
7. Subject is willing and able to provide informed consent to participate or if unable to provide consent have a legal representative who is willing and able to provide informed consent on behalf of the subject.
8. Subject is part of a continence care regimen, defined as "check and change", using any method.
9. If applicable, subject is to be on a stable regimen of medications for urinary incontinence
10. Subject is over 18 years of age.

Exclusion Criteria:

1. Subject has frequent (daily) faecal incontinence in the pad or having severe problems with faecal incontinence as determined by the investigator.
2. Subject has severe incontinence product related skin problems, as defined by the GLOBIAD categorization 2B (skin loss & infection).
3. Subject has any type of indwelling or external urinary catheter(s).
4. Subject is anuric.
5. Subject is managed using another automated or digital health technology incontinence management device.
6. Subject has responsive behaviors of sufficient severity, in the opinion of the care staff, to make participation impractical.
7. Subject has any other condition that makes participation in the clinical investigation inappropriate, as judged by investigator.
8. Subject has a life expectancy of fewer than 3 months or be receiving palliative or terminal care.
9. Subject has participated in an investigational study of a drug, biologic, or device within 30 days prior to entering the clinical investigation or planned during the clinical investigation.
10. Subject is dependent on either alcohol or recreational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Care Efficiency score | 10 weeks.
  Care efficiency is the weighted sum of the pre-defined care events divided by the number of recorded diary days of the subject in question. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily care efficiency score (min/day). Data is collected daily via the study diary.
Daily Skin Health score | 10 weeks.
  Skin health score is based on skin health grades (from 0, no skin problems to 4, very seveer skin problems) that have been reported by the caregiver in the study diary. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily skin health score.

SECONDARY OUTCOMES:
Number of continence care product checks | 10 weeks.
  From the study diary the number of checks of absorbing incontinence products is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of checks.
Number of continence care product changes | 10 weeks.
  From the study diary the number of changes of absorbing incontinence products is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of changes.
Number of continence care toilet visits | 10 weeks.
  From the study diary the number of toilet visits is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of toilet visits.
Number of continence care clothing changes | 10 weeks.
  From the study diary the number of clothing changes due to leakages is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of clothing changes.
Number of continence care bed linen changes | 10 weeks.
  From the study diary the number of bed linen changes due to leakages is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of linen changes.
The time spent on continence care episodes | 10 weeks.
  From the study diary the total time spent on continence care is retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily time spent on continence care.
Skin health score | 10 weeks.
  Measured by the skin health assessment tool at study completion visit and compared to the end of baseline visit.
Quality of life and level of utility | 10 weeks.
  Measured using the EQ-5D-5L questionnaire at study completion visit and compared to the end of baseline visit.
Quality of life according to the QoL-AD | 10 weeks.
  Measured and scored at completion visit and compared to the end of baseline visit.
Level of agitation and responsive behavior. | 10 weeks.
  Measured via interRAI Aggressive Behavior Scale at study completion visit and compared to the end of baseline visit.
Number of sleep interruptions due to continence care | 10 weeks.
  From the study diary the number of sleep interruptions are retrieved. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of interruptions.
Total absorption value | 10 weeks.
  From the study diary the type, number and absorption value of the incontinence care product is retrieved. This data is used to create a total absorption measure. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared.
Caregiver work engagement | 10 weeks.
  Using the UWES questionnaire the work engagement of caregivers are measured at a cluster's end-of-trial visit and compared to the end of baseline visit.
Caregiver work conditions | 10 weeks.
  Measured using the organizational headroom questionnaire at a cluster's end-of-trial visit and compared to the end of baseline visit.
Time spent in a saturated continence care product | 10 weeks
  Data from study diary used to retrieve the total hours that occur between an observed fully saturated product and the change of the saturated product. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily time spent in the saturated product.
Number of unnecessary checks. | 10 weeks
  Data from study diary used to retrieve the number of unnecessary checks/changes. An unnecessary check/change is defined as, an activity line where a product check was performed but no product change occurred or an activity line where a product change occurred but neither a fully nor partially saturated product was indicated. The last week of the 4 week baseline and last week of the 6 week intervention/control time period is to be compared. Data is presented as average daily number of checks/changes.
Qualitative data on implementation, uptake, opportunities and barriers to use. | 10 weeks.
  Response to interviews with caregivers, coded by the investigator and collated into trends and themes. Conducted after completion of study for subjects.
Safety data for the device. | 10 weeks.
  Incidence of adverse events (AE), adverse device effects (ADE), serious adverse events (SAE), serious adverse device effects (SADE), and device deficiency (DD).

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wagg, MD, Principal Investigator — University of Alberta
Locations (2):
- University of Alberta, Edmonton, Alberta, Canada
- Hochschule Niederrhein University of Applied Sciences, Krefeld, Germany